CLINICAL TRIAL: NCT07329842
Title: The Effects of Practitioner Anthropometric Differences and Bed Level on CPR Quality in Pediatric Cardiopulmonary Resuscitation: A Simulation-Based Study
Brief Title: Effect of Bed Height on Chest Compression Quality and Provider Biomechanics During Pediatric CPR Simulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Omür Akınel, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AKDENIZ-PEM-OA-001
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cardiac Arrest (Simulated); Cardiopulmonary Resuscitation, Simulation Training; In-Hospital Cardiac Arrest; Rescuer Fatigue During CPR; CPR Quality Assessment; Bed Height in CPR
Keywords: Cardiopulmonary Resuscitation; CPR Quality; Pediatric Cardiac Arrest; Rescuer Fatigue; Bed Height in CPR

STUDY DESIGN:
Intervention Model Description: Randomized, within-subject 4-condition crossover simulation study. Each participant completes four separate sessions (on different days), performing 2 minutes of single-rescuer, chest-compression-only pediatric CPR per session. Bed height is set to one of four predefined conditions per session; the order of conditions is randomized for each participant.
Masking Description: No masking; bed height condition is apparent to participants and study staff.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fixed Standard Bed Height (58 cm) (Experimental): Participants perform 2 minutes of single-rescuer, chest-compression-only pediatric CPR on a manikin placed on a hospital bed set to a fixed standard height of 58 cm.
  Interventions: Other: Fixed Standard Bed Height (58 cm)
- Anthropometry-Based Bed Height (Patella Midpoint) (Experimental): Participants perform 2 minutes of single-rescuer, chest-compression-only pediatric CPR on a manikin with the hospital bed height adjusted to the participant's patella midpoint (knee midpoint) reference.
  Interventions: Other: Anthropometry-Based Bed Height (Patella Midpoint)
- Anthropometry-Based Bed Height (Lower One-Third of Patella-ASIS Distance) (Experimental): Participants perform 2 minutes of single-rescuer, chest-compression-only pediatric CPR on a manikin with the hospital bed height adjusted to the lower one-third point of the distance between the patella and the anterior superior iliac spine (ASIS).
  Interventions: Other: Anthropometry-Based Bed Height (Lower One-Third Patella-ASIS)
- Self-Selected Bed Height (Experimental): Participants perform 2 minutes of single-rescuer, chest-compression-only pediatric CPR on a manikin with the hospital bed height set to the participant's self-selected "most comfortable/optimal" height.
  Interventions: Other: Self-Selected Bed Height

INTERVENTIONS:
Other: Fixed Standard Bed Height (58 cm) — Hospital bed height is set to a fixed standard height of 58 cm for the CPR session.
  Arms: Fixed Standard Bed Height (58 cm)
Other: Anthropometry-Based Bed Height (Patella Midpoint) — Hospital bed height is adjusted to the participant's patella midpoint reference before the CPR session.
  Arms: Anthropometry-Based Bed Height (Patella Midpoint)
Other: Anthropometry-Based Bed Height (Lower One-Third Patella-ASIS) — Hospital bed height is adjusted to the lower one-third point of the distance between the patella and ASIS before the CPR session.
  Arms: Anthropometry-Based Bed Height (Lower One-Third of Patella-ASIS Distance)
Other: Self-Selected Bed Height — Participant selects the bed height they perceive as optimal/comfortable prior to the CPR session.
  Arms: Self-Selected Bed Height

SUMMARY:
High-quality chest compressions are critical for outcomes after pediatric cardiac arrest, yet rescuer ergonomics and bed height may adversely affect compression quality and fatigue. This randomized crossover simulation study will evaluate how four different bed-height settings influence pediatric CPR quality and rescuer biomechanics. Pediatric emergency medicine residents will perform 2-minute chest-compression-only CPR on a pediatric manikin placed on a hospital bed under four bed-height conditions in randomized order across separate sessions. CPR quality metrics from the manikin's feedback system, rescuer fatigue, physiologic responses, and arm angle over time will be compared to identify an ergonomically optimal bed-height approach.

DETAILED DESCRIPTION:
Background and Rationale

In-hospital pediatric cardiac arrest requires rapid delivery of high-quality CPR. Compression depth, rate, and full chest recoil are key determinants of effective CPR, but maintaining these targets can be challenging due to rescuer posture, bed height, and fatigue. While step-stool use and provider height have been associated with CPR quality in some contexts, there is limited evidence on how bed-height settings-especially anthropometry-based adjustments-affect pediatric CPR performance and rescuer biomechanics over time.

Objective and Hypothesis

Objective: To determine the effect of four bed-height conditions on pediatric CPR quality and rescuer biomechanics in a controlled simulation setting.

Hypothesis: Anthropometry-based and/or self-selected bed height will improve CPR quality (e.g., correct depth and recoil) and reduce perceived exertion compared with a fixed standard bed height.

Study Design

This is a prospective, randomized, within-subject crossover simulation study. Each participant completes CPR under four bed-height conditions, with the order randomized to reduce learning and fatigue bias. Sessions are performed on separate days.

Participants

Eligible participants are volunteer pediatric emergency medicine residents (or comparable clinicians) who are trained in pediatric basic/advanced life support. Individuals with conditions that could limit safe performance of chest compressions (e.g., significant cardiopulmonary or musculoskeletal disorders) are excluded. Anticipated enrollment is approximately 25 participants.

Interventions (Bed-Height Conditions)

Participants will perform chest-compression-only CPR under four bed-height conditions:

Fixed standard bed height (e.g., 58 cm).

Anthropometry-based height A: bed height aligned to a predefined landmark (e.g., patella midpoint).

Anthropometry-based height B: bed height aligned to a second predefined landmark (e.g., a point derived from the distance between patella and anterior superior iliac spine [ASIS]/spina iliaca anterior superior [SIAS], such as the lower one-third point).

Self-selected height: participant chooses the bed height they feel is optimal.

(Replace the anthropometric definitions above with your exact operational definitions.)

Procedures

A pediatric manikin with objective CPR measurement capability (e.g., Laerdal Little Junior QCPR) is placed on a hospital bed. For each condition, the participant performs 2 minutes of continuous chest compressions as a single rescuer. No metronome and no real-time corrective feedback are provided during the compression period (unless your protocol uses feedback; then adjust this sentence). Standardized hand placement and compression position are instructed.

Outcome Measures

Primary Outcome

Correct Compression Depth (%) during each 2-minute session (manikin-derived).

Secondary Outcomes

Average compression depth (mm)

Average compression rate (compressions/min)

Correct chest recoil / release (%)

Composite CPR quality scores (e.g., compression score, total score), as available from the manikin system

Rescuer fatigue: Borg Rating of Perceived Exertion immediately after each session

Physiologic response: heart rate and oxygen saturation (SpO₂) measured pre- and post-session (and change from baseline)

Rescuer biomechanics: arm/upper-limb angle measured from video at standardized time points during compressions (e.g., 0, 30, 60, 90, 120 seconds)

Statistical Considerations

Outcomes will be compared across bed-height conditions using within-subject methods (e.g., linear mixed-effects models with participant as a random effect). Pairwise comparisons will be adjusted for multiple testing. Exploratory analyses may evaluate whether participant anthropometry (height, BMI, etc.) modifies the effect of bed height on CPR quality.

Ethical Considerations

This is a simulation-based study with no patient involvement and minimal risk. Participants may stop at any time due to discomfort or fatigue. The study has ethics approval from [Akdeniz Üniversitesi Bilimsel Araştırma ve Yayın Etiği Kurulu, Approval Number: 875 /09/28/2025] and all participants provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pediatric resident/assistant physician working in the Department of Pediatrics (Akdeniz University) with valid ÇİYAD certification
* Willing and able to provide written informed consent
* Able to perform a 2-minute continuous chest-compression CPR cycle on a pediatric manikin
* Available to complete four CPR sessions (each at a different bed-height condition) on separate days

Exclusion Criteria:

* Known chronic cardiopulmonary disease that may limit physical exertion during CPR
* Known musculoskeletal disorder or chronic condition that may affect CPR performance
* Acute injury/illness at the time of participation that could impair safe CPR performance
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Correct chest compression depth (%, QCPR-defined) | During each 2-minute chest compression-only CPR session (per bed-height condition).
  Percentage of compressions meeting the target depth criteria as calculated by Laerdal Little Junior QCPR manikin sensors. (Recorded separately for each bed-height condition.)

SECONDARY OUTCOMES:
Average chest compression depth (mm) | During each 2-minute chest compression-only CPR session (per bed-height condition).
  Mean compression depth (mm) recorded by the QCPR manikin.
Average chest compression rate (compressions/min) | During each 2-minute chest compression-only CPR session (per bed-height condition).
  Mean compression rate (compressions/min) recorded by the QCPR manikin.
Correct chest recoil / release (%, QCPR-defined) | During each 2-minute chest compression-only CPR session (per bed-height condition).
  ercentage of compressions with complete release (recoil) as calculated by the QCPR manikin.
Perceived exertion (Borg RPE score) | Immediately after each 2-minute CPR session.
  Borg scale score collected verbally at the end of each CPR cycle.
Change in heart rate (beats/min) | From immediately before to immediately after each 2-minute CPR session.
  Post-CPR heart rate minus pre-CPR heart rate measured by pulse oximeter.
Change in oxygen saturation (SpO2, %) | From immediately before to immediately after each 2-minute CPR session.
  Post-CPR SpO2 minus pre-CPR SpO2 measured by pulse oximeter.
Arm angle during CPR (degrees) | During each 2-minute CPR session (0, 30, 60, 90, and 120 seconds).
  Arm/trunk angle measured from standardized video frames captured at 0, 30, 60, 90, and 120 seconds; angle derived via software-based measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital / Faculty of Medicine Hospital - Dept. of Pediatrics, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No